CLINICAL TRIAL: NCT01832623
Title: Are Bone, Nutritional and Cardiovascular Status of French Children and Adolescents, Correlated With Their Vitamin D Status?
Brief Title: Vitamin D, Bones, Nutritional and Cardiovascular Status
Acronym: VITADOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011.688
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2017-02

CONDITIONS: Vitamin D
Keywords: Vitamin D; bone; cardiovascular status; nutritional status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exploration of Vitamin D roles (Experimental): Various exams will be performed during two visits (the same day or within three months) in order to answer the objectives of the study.
  Interventions: Other: Exploration of Vitamin D roles

INTERVENTIONS:
Other: Exploration of Vitamin D roles — * Visit 1: questioning, physical examination, blood sampling (including plasma collection for future genetic analyses), carotid ultrasound
  * Visit 2 (same day as visit 1 or maxi 3 months later): HR-pQCT, dual energy x-ray absorptiometry (DXA), iontophoresis of acetylcholine and sodium nitroprusside

SUMMARY:
Vitamin D is not seen anymore only as a phosphocalcic hormone, but also as having an effect on global health (anti-infective, anti-inflammatory, anti-tumour roles and cardiovascular protection).

The link between vitamin D deficiency and osteomalacia lesions is well-known. In paediatrics, systematic vitamin D supplementation of infants and toddlers, associated with milk enrichment, has allowed an almost total disappearance of rickets. Vitamin D repletion was defined as the minimal concentration that enables the prevention of rickets in children and osteomalacia in adults, that is approximately 8 ng/mL (20 nmol/L). However, in 2010, most of the international experts agreed to set minimal threshold of 25 OH vitamin D serum concentration, higher than the one previously admitted, with a limit of 20 ng/mL (50 nmol/L) to define a vitamin D deficiency and a limit of 30 ng/mL (75 nmol/L) to define vitamin D insufficiency in adults. In the paediatric population, the consensus is less obvious and we consider that a serum concentration of minimum 20 ng/mL is necessary.

A study on more than 200 children from Lyon, followed in the paediatric nephrology unit and having a renal function normal or sub-normal, demonstrated an important prevalence of vitamin D deficiency (75%) in adolescents and pre-adolescents.

Concurrently, the appearance of new bone imaging techniques (especially high-resolution peripheral quantitative computed tomography HR-pQCT) improved bone status evaluation in a non-invasive manner.

Given the new pathophysiological data on pleiotropic role of vitamin D (bone, cardiovascular system, adipose tissue) and given the proportion of French children possibly suffering from vitamin D deficiency, it seems urgent to actualize current recommendations regarding systematic supplementation in vitamin D. This transversal study on 200 healthy children and adolescents will allow to have an overview of vitamin D status in French healthy children and adolescents, studying with non-invasive, safe, reliable and innovative tools, the theoretical targets of vitamin D (bones, cardiovascular system and nutritional status); and then to lay the foundations of therapeutic trials aiming to evaluate the mode of vitamin D supplementation for healthy children and adolescents; while having a cohort for HR-pQCT measurements, that will allow us to have French reference range in a 10-17 year-old population, for this innovative, non-invasive and low radiation exposure technique.

DETAILED DESCRIPTION:
To study the correlation between bone assessment by high-resolution peripheral quantitative computed tomography (HR-pQCT) and vitamin D serum concentration.

ELIGIBILITY:
Inclusion Criteria:

* 10 year-old <or= Age < 18 year-old
* Without mobility handicap (medical walker, crutch, wheelchair…)
* Written informed consent (signed by parents)

Exclusion Criteria:

* History of treatment with growth hormone
* History of treatment with oral corticoids, taken over more than 3 consecutive months
* Current treatment with growth hormone, corticoids or anti-calcineurin
* Treatment with aspirin or nonsteroidal anti-inflammatory drug within the last three weeks
* Treatment with paracetamol within the last week
* Chronic pathology with an impact on growth:

  * Parenteral nutrition
  * Chronic inflammatory disease (rheumatologic or digestive notably)
  * System diseases (lupus, granulomatosis, vascularitis)
  * Renal failure
  * Diabetes
* Serious intercurrent disease (infection, neoplasia)
* Ongoing pregnancy
* Patient unaffiliated with the French universal healthcare system.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To study the correlation between the results of bone microarchitecture obtained by high-resolution peripheral quantitative computed tomography (HR-pQCT) and vitamin D serum concentration. | up to 3 months
  The HR-pQCT evaluates bones down to the level of the tiny individual elements that nature configures in a way that makes bones as strong as possible. HR-pQCT measures bone density and quantifies the three dimensional geometry, strength and microarchitecture of bone at the lower arm (radius) and lower leg (tibia).

SECONDARY OUTCOMES:
Values and standard deviation of 25-OH vitamin D3 plasma concentration concentration in the population studied. | Once. At inclusion (V1).
  Blood intake.
To study the correlation between vitamin D plasma concentration and nutritional and pubertal status, cardiovascular status, inflammatory status . | up to 3 months
  Nutritional and pubertal status will be assessed thanks to: Body Mass Index, Dual-energy X-ray Absorptiometry, adipokines level. Cardiovascular status will be assessed thanks to arterial pressure, Intima-media Thickness (IMT), Extra-media Thickness (EMT), lipid profile, endothelial function. IMT and EMT will be obtained using carotid ultrasound. Endothelial function will be evaluated following a protocol of iontophoresis of acetylcholine and sodium nitroprusside.
  Inflammatory status will be measured looking at C-reactive protein plasma level.
To evaluate the relation between bone parameters (HR-pQCT) and adipokines; and the relation between bone parameters and cardio-vascular data (blood pressure, IMT, EMT, lipid profile, endothelial function). | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bachetta, MD, Principal Investigator — Centre de Référence des Maladies Rénales Rares - Hospices Civils de Lyon - Service de Néphrologie et Rhumatologie Pédiatriques - Hôpital Femme Mère Enfant - 69500 BRON - FRANCE
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, France

REFERENCES:
- [Result] Preka E, Ranchin B, Doyon A, Vierge M, Ginhoux T, Kassai B, Bacchetta J. The interplay between bone and vessels in pediatric CKD: lessons from a single-center study. Pediatr Nephrol. 2018 Sep;33(9):1565-1575. doi: 10.1007/s00467-018-3978-3. Epub 2018 Jun 5. PMID 29872964